CLINICAL TRIAL: NCT06282380
Title: Fibricheck Detection cApabilities for Atrial Fibrillation - a Multicenter Validation Study
Brief Title: Fibricheck Detection cApabilities for Atrial Fibrillation
Acronym: FDA-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qompium NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FDA-AF study
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- FibriCheck Mobile Application measurements (Other): Participants will perform one measurement using the FibriCheck Mobile Application and the result will be compared with the ground truth.
  Interventions: Device: FibriCheck Mobile Application

INTERVENTIONS:
Device: FibriCheck Mobile Application — PPG measurement with reference diagnosis

SUMMARY:
Evaluation of accuracy of the FibriCheck Mobile Application on various smartphone devices, compared to the reference diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* At least 22 years old;
* Capable of independently performing FibriCheck recordings (researcher-observed);
* Cardiology patients, hospitalized/in-clinic or consulting the cardiac outpatient clinic, with or without a diagnosis of atrial fibrillation.

Exclusion Criteria:

* Individuals with cardiac pacemakers, implantable cardioverter-defibrillators, or other implanted electronic devices as these can influence the natural heart rhythm;
* Individuals enrolled in another clinical trial;
* Individuals with physical or medical characteristics that prevent them from successfully taking a measurement e.g. extreme callus (i.e., rough or thickened area of skin fingertip), tremor, cognitive impairment, Parkinson's disease;
* Pregnant and/or nursing women.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Accuracy of the FibriCheck Mobile Application | Through study completion: 1 day
  Accuracy based on the reference diagnosis

SECONDARY OUTCOMES:
Sensitivity of the FibriCheck Mobile Application | Through study completion: 1 day
  Sensitivity based on the reference diagnosis
Specificity of the FibriCheck Mobile Application | Through study completion: 1 day
  Specificity based on the reference diagnosis

CONTACTS AND LOCATIONS:
Locations (5):
- United States (3):
  - Northwestern Medicin, Chicago, Illinois
  - New York Presebyterian Queens, New York, New York
  - OU Medicine College, Oklahoma City, Oklahoma
- Belgium (2):
  - University Hospital Antwerp, Antwerp
  - Ziekenhuis Oost-Limburg, Genk

IPD SHARING:
Plan to Share IPD: No